CLINICAL TRIAL: NCT00428610
Title: A Phase 2 Study of LY573636-Sodium as Treatment for Patients With Platinum-Resistant Ovarian Cancer
Brief Title: A Study of Chemotherapy Treatment for Patients With Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10410; H8K-MC-JZAG (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-01-26; First posted 2007-01-30 (Estimated); Results first posted 2018-04-19 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-03

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — N-((5-bromo-2-thienyl)sulfonyl)-2,4-dichlorobenzamide

ARMS (1):
- LY573636 (Experimental): LY573636-sodium (LY573636) is administered every 28 days until disease progression or other criteria for participant discontinuation are met.
  Interventions: Drug: LY573636-sodium

INTERVENTIONS:
Drug: LY573636-sodium — LY573636 dose is dependent on participant's height, weight, and gender and is adjusted to target a specific maximum concentration (Cmax) based on participant laboratory parameters. LY573636 is administered every 28 days until disease progression or other criteria for participant discontinuation are met.
  Other Names: tasisulam; LY573636

SUMMARY:
The primary objective is to determine whether LY573636-sodium (hereafter referred to as LY573636) is effective in treating platinum-resistant ovarian cancer. Patients will receive an intravenous infusion of study drug once every 28 days. Computed tomography (CT) scans and CA-125 tests will be done before the first dose and then after every other treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer
* At least 18 years old
* Have received at least one but no more than 2 systemic treatment regimens containing platinum (does not include regimens received before surgery for this cancer)
* Have platinum-resistant disease

Exclusion Criteria:

* Have received more than 2 systemic treatment regimens for platinum-resistant disease
* Serious pre-existing medical conditions
* Actively receiving warfarin (Coumadin) for treatment of venous thrombosis or other prothrombotic conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2007-02; Primary Completion 2011-02 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
- Italy (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brescia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow, Russia

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The reasons for discontinuation listed in the participant flow are the reasons the participant discontinued treatment and a participant was considered to have "completed" the trial if they experienced progressive disease or an adverse event.
Groups:
- Target Cmax 420 µg/mL: Loading dose of LY573636, targeting a maximum concentration (Cmax) of 420 micrograms/milliliter (μg/mL), followed by a lower chronic dose (which was 75% of the loading dose) in subsequent cycles, administered as an intravenous infusion given over approximately 2 hours, on Day 1 of a 21-day treatment cycle.
- Target Cmax 360 μg/mL: Loading dose of LY573636, targeting a Cmax of 360 μg/mL, followed by a lower chronic dose (which was 90% of the loading dose) in subsequent cycles, administered as an intravenous infusion given over approximately 2 hours, on Day 1 of a 21-day treatment cycle.
- Albumin-Tailored Dose: The dose of LY573636 administered in each infusion was based on participant's height, weight, gender, pre-cycle albumin level, and cycle number to target area under the curve above the albumin corrected threshold (AUCalb) in the range of 1200 to 6400 hour*micrograms/milliliter (h*μg/mL), administered over approximately 2 hours on Day 1 of a 28-day treatment cycle.
Period: Overall Study
Arm/Group | Target Cmax 420 µg/mL | Target Cmax 360 μg/mL | Albumin-Tailored Dose
Started | 53 | 18 | 32
Received at Least One Dose of Study Drug | 53 | 18 | 32
Completed | 0 | 0 | 0
Not Completed | 53 | 18 | 32
Not completed — Death Due to Adverse Event | 3 | 0 | 5
Not completed — Death Due to Progressive Disease | 0 | 0 | 2
Not completed — Adverse Event | 2 | 3 | 2
Not completed — Investigator Decision | 2 | 1 | 1
Not completed — Progressive Disease | 42 | 14 | 22
Not completed — Withdrawal by Subject | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who had at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Target Cmax 420 µg/mL | Target Cmax 360 μg/mL | Albumin-Tailored Dose | Total
Number analyzed (Participants) | 53 | 18 | 32 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.88 (11.12) | 59.88 (8.98) | 56.83 (10.37) | 57.39 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 18 | 32 | 103
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Decent (black) | 1 | 0 | 1 | 2
  Caucasian | 50 | 18 | 31 | 99
  East Asian | 1 | 0 | 0 | 1
  Hispanic | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 10 | 21 | 63
  Russia | 12 | 0 | 0 | 12
  Italy | 9 | 8 | 11 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response and Partial Response (Objective Response Rate)
Description: Objective response is complete response (CR) + partial response (PR), as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines. CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions. Objective response rate is calculated as a total number of participants with CR or PR divided by the total number of participants treated multiplied by 100.
Time Frame: Baseline to measured progressive disease up to 12.68 months
Population: All participants who received at least one dose of the study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Target Cmax 420 µg/mL | Target Cmax 360 μg/mL | Albumin-Tailored Dose
Number analyzed (Participants) | 53 | 18 | 32
percentage of participants | 7.5 [1.6 to 13.5] | 0 [NA to NA] — No participant had CR or PR, therefore 90% Confidence Interval was not calculable. | 3.1 [0.0 to 8.2]

2. Secondary Outcome: Progression Free Survival
Description: Defined as the time from date of first dose to the first observation of progression of disease (PD) or death due to any cause. PD was determined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. PD is ≥20% increase in sum of longest diameter of target lesions and/or a new lesion.
Time Frame: Baseline to measured progressive disease or death due to any cause up to 21.26 months
Population: All participants who received at least 1 dose of the study drug.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Target Cmax 420 µg/mL | Target Cmax 360 μg/mL | Albumin-Tailored Dose
Number analyzed (Participants) | 53 | 18 | 32
months | 1.87 [1.41 to 3.02] | 2.40 [1.61 to 3.35] | 2.10 [1.87 to 3.22]

3. Secondary Outcome: Percentage of Participants With Complete Response, Partial Response, and Stable Disease (Clinical Benefit Rate)
Description: Clinical Benefit Rate is complete response (CR) + partial response (PR) + stable disease (SD) as classified by the investigator according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines. CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. Clinical benefit rate is calculated as a total number of participants with CR or PR or SD divided by the total number of participants treated multiplied by 100.
Time Frame: Baseline to measured progressive disease up to 21.26 months
Population: All participants who received at least one dose of the study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Target Cmax 420 µg/mL | Target Cmax 360 μg/mL | Albumin-Tailored Dose
Number analyzed (Participants) | 53 | 18 | 32
percentage of participants | 45.3 [34.0 to 56.5] | 61.1 [42.2 to 80.0] | 34.4 [20.6 to 48.2]

4. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY573636
Time Frame: Predose up to 2 hours postdose in Cycles 1 and 2
Population: All participants who received at least one dose of the study drug and had pharmacokinetics data at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (µg/mL)
Arm/Group | Target Cmax 420 µg/mL | Target Cmax 360 μg/mL | Albumin-Tailored Dose
Number analyzed (Participants) | 51 | 17 | 32
micrograms/milliliter (µg/mL)
  Cycle 1 | 368.4 (8.9) | 324.1 (7.9) | 340.9 (15.4)
  Cycle 2: number analyzed (Participants) | 45 | 16 | 29
  Cycle 2 | 323.0 (13.6) | 326.1 (14.5) | 320.7 (17.7)

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from date of first treatment to the date of death due to any cause. For participants who were alive, overall survival was censored at their last contact.
Time Frame: First treatment to death due to any cause up to 42.91 months
Population: All participants who received at least one dose of the study drug. The numbers of participants censored are 11 (Target Cmax 420 µg/mL group), 6 (Target Cmax 360 µg/mL group) and 14 (Albumin-Tailored Dose group).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Target Cmax 420 µg/mL | Target Cmax 360 μg/mL | Albumin-Tailored Dose
Number analyzed (Participants) | 53 | 18 | 32
months | 13.08 [7.66 to 21.36] | 10.09 [8.02 to 22.97] | 11.63 [7.20 to NA] — The upper limit of the 90% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

6. Secondary Outcome: Duration of Response
Description: The duration of response (complete response [CR] or partial response [PR]) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause. CR or PR is classified by the investigators according to Response Evaluation Criteria In Solid Tumors (RECIST) guidelines. CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions.
Time Frame: Time of response to time of measured progressive disease up to 12.68 months
Population: All participants who received at least one dose of the study drug and had complete response (CR) or partial response (PR).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Target Cmax 420 µg/mL | Target Cmax 360 μg/mL | Albumin-Tailored Dose
Number analyzed (Participants) | 4 | 0 | 1
months | 5.03 [2.99 to 6.21] |  | 12.68 [NA to NA] — Only 1 participant had PR, therefore 90% Confidence Interval was not calculable.

7. Secondary Outcome: Duration of Stable Disease
Description: Duration of stable disease is defined from date of documented stable disease (SD) or better to first date of progressive disease or death from any cause (assessed every cycle during study therapy, or every 2 months during post-therapy until disease progression or death). SD is neither sufficient shrinkage to qualify for partial response (PR) nor sufficient increase to qualify for PD. PR is ≥30% decrease in sum of longest diameter of target lesions. PD is ≥20% increase in sum of longest diameter of target lesions and/or a new lesion.
Time Frame: Time from documented SD or better to first date of progressive disease or death due to any cause up to 21.26 months
Population: All participants who received at least one dose of the study drug and stable disease or better.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Target Cmax 420 µg/mL | Target Cmax 360 μg/mL | Albumin-Tailored Dose
Number analyzed (Participants) | 24 | 11 | 11
months | 3.71 [2.76 to 4.21] | 3.27 [2.79 to 10.02] | 3.78 [3.22 to 5.59]

8. Secondary Outcome: Number of Participants With Adverse Events (Safety)
Description: Data are presented as number of participants who experienced serious adverse events or all other nonserious adverse events during the study including the 30-day follow-up period. A summary of serious adverse events and other nonserious adverse events is located in the Reported Adverse Event section.
Time Frame: First treatment dose up to 43.91 months
Population: All participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Target Cmax 420 µg/mL | Target Cmax 360 μg/mL | Albumin-Tailored Dose
Number analyzed (Participants) | 53 | 18 | 32
Participants
  Serious Adverse Events | 21 | 5 | 15
  Other Nonserious Adverse Events | 47 | 18 | 30

9. Other Pre Specified Outcome: Number of Participants Who Died Due to Progressive Disease During the 30 Days Following Discontinuation From Study Treatment
Time Frame: Study treatment discontinuation up to 30 days post study treatment discontinuation
Population: All participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Target Cmax 420 µg/mL | Target Cmax 360 μg/mL | Albumin-Tailored Dose
Number analyzed (Participants) | 53 | 18 | 32
Participants | 2 | 3 | 1

ADVERSE EVENTS:
Description: Deaths due to progressive disease are not considered adverse events; however they are reported in the participant flow for those who died during the study and in the Other Pre-Specified outcome measure for those who died during the 30-day post study treatment follow-up period.
Arm/Group | Target Cmax 420 µg/mL | Target Cmax 360 μg/mL | Albumin-Tailored Dose
Serious Adverse Events (participants affected / at risk) | 21/53 | 5/18 | 15/32
Other Adverse Events (participants affected / at risk) | 47/53 | 18/18 | 30/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Target Cmax 420 µg/mL (N=53) | Target Cmax 360 μg/mL (N=18) | Albumin-Tailored Dose (N=32)
Anaemia (Blood and lymphatic system disorders) | 5 (7) | 2 (2) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7) | 2 (2) | 7 (7) — Resulted in 1 death in the Albumin-Tailored Dose arm.
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Resulted in 1 death in the Albumin-Tailored Dose arm.
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Resulted in 1 death in the Target Cmax 420 µg/mL arm.
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) — Resulted in 1 death in the Target Cmax 420 µg/mL arm.
Intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 1 (1) | 3 (3)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Resulted in 1 death in the Target Cmax 420 µg/mL arm within 30 days of discontinuation from study treatment.
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 1 (1) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0) | 2 (2)
Hyperpyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess intestinal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Resulted in 1 death in the Albumin-Tailored Dose arm.
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 1 (2) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) — Resulted in 1 death in the Target Cmax 420 µg/mL arm.
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Resulted in 1 death in the Target Cmax 420 µg/mL arm within 30 days of discontinuation from study treatment.
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Resulted in 1 death in the Albumin-Tailored Dose arm.
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) — Resulted in 1 death in the Albumin-Tailored Dose arm.
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Target Cmax 420 µg/mL (N=53) | Target Cmax 360 μg/mL (N=18) | Albumin-Tailored Dose (N=32)
Anaemia (Blood and lymphatic system disorders) | 10 (13) | 5 (6) | 4 (5)
Leukopenia (Blood and lymphatic system disorders) | 4 (7) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 12 (17) | 2 (2) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 18 (28) | 4 (5) | 3 (4)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 4 (4) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 10 (12) | 1 (1) | 5 (5)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 7 (7) | 2 (2) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 12 (17) | 7 (10) | 7 (8)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 1 (1) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 16 (20) | 4 (5) | 12 (14)
Stomatitis (Gastrointestinal disorders) | 6 (8) | 2 (3) | 7 (7)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 4 (4) | 7 (8)
Asthenia (General disorders) | 2 (2) | 4 (4) | 7 (7)
Chills (General disorders) | 0 (0) | 2 (2) | 1 (1)
Early satiety (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 25 (43) | 5 (5) | 4 (4)
Injection site pain (General disorders) | 2 (2) | 1 (1) | 2 (2)
Malaise (General disorders) | 1 (1) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 2 (2) | 1 (1)
Pain (General disorders) | 3 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 2 (2) | 2 (3)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear lobe infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 4 (4) | 1 (1) | 3 (3)
Influenza (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 3 (5) | 1 (2)
Body temperature (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1) | 4 (4)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 3 (3)
Weight decreased (Investigations) | 3 (3) | 0 (0) | 3 (3)
Weight increased (Investigations) | 2 (3) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 2 (4)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 6 (8)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (8) | 2 (2) | 5 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 8 (8) | 1 (1) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 4 (4) | 3 (4)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 6 (6) | 2 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 3 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 5 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10) | 0 (0) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 14 (25) | 0 (0) | 3 (4)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days